CLINICAL TRIAL: NCT01416207
Title: A Multiple-Dose, Open-Label, Phase 1, Pharmacokinetic, Pharmacodynamic, and Safety Study of Avonex® in Chinese Healthy Volunteer Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Biogen Idec Limited
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 108HV105
Record Dates: First submitted 2011-06-30; First posted 2011-08-12 (Estimated); Last update posted 2011-11-04 (Estimated); Status verified 2011-11

CONDITIONS: Healthy
MeSH Terms: interventions — Interferon beta-1a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Avonex (Experimental): 4 weekly injections of Avonex (IM)
  Interventions: Drug: Avonex

INTERVENTIONS:
Drug: Avonex — 4 weekly injections of Avonex (IM)
  Other Names: Interferon-β1a

SUMMARY:
Rationale for the Study:

The purpose of this study is to characterize the pharmacokinetic (PK) and pharmacodynamic (PD) profile of Avonex in Chinese healthy volunteer subjects. Data from this study will be used to support registration of Avonex in China.

Study Design:

This is a multiple-dose, single-arm, open-label, PK/PD and safety study. Four weekly injections of Avonex will be administered intramuscularly (IM). Frequent (intensive) blood samples will be collected with the first and fourth injections of Avonex, and a sparse blood sample will be collected with the second and third injections of Avonex.

DETAILED DESCRIPTION:
Rationale for the Study:

The purpose of this study is to characterize the pharmacokinetic (PK) and pharmacodynamic (PD) profile of Avonex in Chinese healthy volunteer subjects. Data from this study will be used to support registration of Avonex in China.

Study Design:

This is a multiple-dose, single-arm, open-label, PK/PD and safety study. Four weekly injections of Avonex will be administered intramuscularly (IM). Frequent (intensive) blood samples will be collected with the first and fourth injections of Avonex, and a sparse blood sample will be collected with the second and third injections of Avonex.

Four Avonex IM injections will be administered in this study. Due to the long-term use of Avonex by MS patients, a multiple-dose PK/PD study is necessary in order to provide adequate information to evaluate changes in drug concentrations over time in Chinese healthy subjects. Serum levels of interferon beta in Caucasian healthy volunteers have been shown to peak between 3 and 15 hours after administration of Avonex IM at the dose being used in this study and have been shown to decline at a rate consistent with a 10-hour elimination half-life; therefore, accumulation of interferon beta following multiple weekly Avonex IM injections is not anticipated.

Exposure of healthy subjects to multiple doses of Avonex in this study is not anticipated to present safety or tolerability issues based on experience from previous Avonex studies that have been conducted in healthy volunteer subjects and MS patients. Flu-like symptoms associated with this dose of Avonex have generally been mostly of mild-to-moderate intensity and of short duration, typically experienced within the first 24 hours after injection. Prophylactic analgesic medication must be administered prior to each Avonex injection during the study which is a recommended practice with the use of interferon therapies in order to ameliorate flu-like symptoms.

Study Location:

China, at 1 Phase 1 study site.

Duration of Treatment and Follow-up:

Approximately 2 months, including a 28-day Screening and Baseline period, a 3-week Treatment and blood sampling period and a 14-day Follow-Up period.

Statistical Methods:

PK/PD parameters will be calculated using non-compartmental methods. Summary statistics for each PK/PD parameter will be calculated. Mean concentration values will be plotted over time both on a linear and a logarithmic scale.

The incidence of treatment-emergent AEs will be summarized. Vital signs will be examined to determine the incidence of clinically relevant abnormalities.

Laboratory evaluations will be assessed to determine the incidence of abnormalities. Changes in laboratory evaluations will be summarized using shift tables and summary statistics.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations.
* Subjects of Chinese origin (at least both maternal and paternal grandparents of Chinese origin).
* Body mass index (BMI) within the range of 18.5 to 30 kg/m2 (inclusive).
* All male subjects and female subjects of childbearing potential must practice effective contraception during the study and be willing and able to continue contraception for 30 days after their last dose of study treatment.

Exclusion Criteria:

* History of seizure disorder or unexplained blackouts OR history of a seizure within 6 months prior to Day 1.
* History of suicidal ideation or an episode of clinically severe depression (as determined by the Investigator) within 6 months prior to Day 1.
* Any clinically significant presence (as determined by the Investigator) of cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, or other major disease.
* Positive test result for hepatitis C antibody (HCV Ab), or current hepatitis B infection at Screening.
* Known history of human immunodeficiency virus (HIV).
* Clinically significant abnormal laboratory values.
* History of alcohol abuse (as defined by the Investigator), or a positive blood screen test for presence for alcohol at Screening.
* History of drug abuse (as defined by the Investigator), or a positive urinary screen test for presence of cocaine and morphine.
* Premalignant and malignant disease.
* History of clinically significant severe allergic or anaphylactic reactions.
* Known allergy to any component of the Avonex formulation.
* History of hypersensitivity or intolerance to prophylactic analgesic medication that would preclude use during the study.
* Clinically significant abnormal electrocardiogram (ECG) values as determined by the Investigator.
* Known allergy to interferon beta-1a.
* Active bacterial or viral infection.
* Female subjects who are pregnant or currently breastfeeding.
* Previous participation in another investigational drug study within the last 1 month or 7 half-lives, whichever is longer, or previous participation in this study.
* Treatment with any prescription medication within 14 days of Day 1.
* Treatment with any over-the-counter products within the 14 days prior to Day 1.
* Donation of blood (500 mL or greater) within 56 days prior to Day 1.
* Inability to comply with study requirements

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Cmax | Participants will be followed for the duration of the study; and expected 2 months
Tmax | Participants will be followed for the duration of the study; and expected 2 months
AUC 0-t | Participants will be followed for the duration of the study; and expected 2 months
AUC 0-infinity | Participants will be followed for the duration of the study; and expected 2 months
T 1/2 | Participants will be followed for the duration of the study; and expected 2 months
Tlag | Participants will be followed for the duration of the study; and expected 2 months
Ka | Participants will be followed for the duration of the study; and expected 2 months
T 1/2ab | Participants will be followed for the duration of the study; and expected 2 months
Kcl | Participants will be followed for the duration of the study; and expected 2 months
Kir | Participants will be followed for the duration of the study; and expected 2 months
Emax | Participants will be followed for the duration of the study; and expected 2 months
Tmax(E) | Participants will be followed for the duration of the study; and expected 2 months
Eauc | Participants will be followed for the duration of the study; and expected 2 months
Induction ratio | Participants will be followed for the duration of the study; and expected 2 months
T1/2 return to baseline | Participants will be followed for the duration of the study; and expected 2 months

SECONDARY OUTCOMES:
Number of Adverse Events as a measure of safety and tolerability | Participants will be followed for the duration of the study; and expected 2 months
Number of Serious Adverse Events as a measure of safety and tolerability | Participants will be followed for the duration of the study; and expected 2 months
Changes in lab assessments | Participants will be followed for the duration of the study; and expected 2 months
Changes in vital signs | Participants will be followed for the duration of the study; and expected 2 months
Changes in physical examinations | Participants will be followed for the duration of the study; and expected 2 months
Changes in ECGs | Participants will be followed for the duration of the study; and expected 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Shanghai, China